CLINICAL TRIAL: NCT03980899
Title: Valuation of the Long-term Tolerance of Proton Pump Inhibitor (PPI) Discontinuation in Geriatric Patients Treated With Long-term Therapy Without a Recognized Indication
Brief Title: Evaluation of the Long-term Tolerance of Proton Pump Inhibitor (PPI) Discontinuation in Geriatric Patients Treated With Long-term Therapy Without a Recognized Indication
Acronym: EGERIPP 2
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EGERIPP 2
Record Dates: First submitted 2019-06-07; First posted 2019-06-10 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Proton Pump Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PPI

SUMMARY:
Proton pump inhibitors (PPIs) are widely prescribed in France as anti-ulcer drugs. The indications currently approved in France, with variations according to molecules, are as follows: eradication of Helicobacter pylori, active peptic ulcer disease, maintenance treatment of duodenal ulcer disease, treatment of gastroduodenal lesions induced by non-steroidal anti-inflammatory drugs (NSAIDs), prevention of NSAID-induced gastro-duodenal lesions in at-risk subjects, symptomatic treatment of gastroesophageal reflux disease (GERD), esophagitis by GERD, maintenance treatment of esophagitis by GERD and Zollinger-Ellison syndrome.

Several misuse situations had been identified by the High Authority of Health (HAS) in its reassessment in 2009.

Although these molecules are very well tolerated in the short term, studies show the occurrence of long-term adverse effects such as an increase in the number of lung infections, Clostridium difficile infections and an increased risk of fractures.

DETAILED DESCRIPTION:
Professor Sylvie Legrain, in a 2005 HAS report, described that "Better prescribing in the elderly is thus a public health issue. "Indeed, although multi-medication in the elderly is often justified, it increases the risk of drug iatrogeny, reduces compliance and has a significant cost to society. In this report, it is specified that digestive tract drugs (including PPIs) represent the 3rd most prescribed class of drugs for people over 65 years of age (17% of patients use them regularly). PPIs are also mentioned in this report as overuse (overtreatment).

The first study, conducted in 2017 at our centre (EGERIPP), sought to assess whether a rebound effect was observed in patients who stopped PPI therapy (if not indicated). In this study, 30 patients were included and no rebound effects were observed. Five patients resumed PPIs out of the 30 patients included (unexplored anemia - n=1, epigastric pain - n=1, gastroesophageal reflux disease - n=1, no justification found - n=2). For all patients, during reassessment on D14 and D21 (during hospitalization), patients did not report more symptoms after discontinuation. In this context, the investigators now wish to study whether the short-term tolerance is prolonged in the long term for the discontinuation of PPIs.

This first study also allowed us to assess the prevalence of PPI use in the elderly, and the prevalence of patients on PPI for a recognized indication. During the study, 270 patients were screened and 76 patients had a PPI at admission (28%). Of these 76 patients, no indication recognized by the HAS was found in the medical file for 63 patients (83%).

The discontinuation of PPI treatments in case of use outside the recommendations is usually carried out in the department where the study is being conducted. There is therefore no change in practices. On the other hand, it is good practice to discontinue a treatment that is prescribed outside the recommendations.

Following the EGERIPP study, the systematic reassessment of PPI treatments has become a service practice, with discontinuation when no recognized indication is found and prescription of antacids on demand.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in post acute and rehabilitation service
* more than 65 years old
* French-speaking patient
* Patients with PPI* in their SSRG entry treatment in an indication not recognized by the HAS and which has therefore been stopped (according to the service protocol)

Exclusion Criteria :

* Patient with a justified indication of PPI (recognized by the HAS)
* Patient receiving an IVSE PPI (pantoprazole 8mg/h) for suspected GI bleeding, even if not proven.
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under the protection of justice
* Patient opposing participation in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient admitted in Leopold Bellan post acute an rehabilitation institution.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with one or more of symptoms at Month 3 | 3 months after end of treatment
  Percentage of patients with one or more of the following symptoms at Month 3 after PPI discontinuation: dyspepsia, reflux, heartburn, persistent dry cough, gastralgia (symptoms expected when PPI discontinuation occurs)

SECONDARY OUTCOMES:
Percentage of patients who have experienced one or more symptoms | 14 days after end of treatment
  Percentage of patients who have experienced one or more of the following symptoms since stopping: dyspepsia, reflux, heartburn, persistent dry cough and/or gastralgia.
Cumulative number of antacid intakes within 14 days of stopping PPIs | 14 days after end of treatment
Comparaison of percentage | Day 14 and Month 3
  comparison of the:
  * Percentage of patients who experienced at least one of the above symptoms
  * Percentage of patients who felt they had experienced more of these symptoms
Proportion of patients who resumed PPI treatment and reason for resumption | Day 14 and Month 3
Proportion of patients for whom the use of PPIs and their drug treatments in general is "very high" or "very important" | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Bernard P DURAND GASSELIN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France